CLINICAL TRIAL: NCT00631488
Title: A Phase IIa, Multicenter, Double-Blind, Randomized, Active Comparator-Controlled Clinical Trial to Study the Efficacy and Safety of MK0893 in Combination With Sitagliptin or in Combination With Metformin in Patients With Type 2 Diabetes Mellitus Who Have Inadequate Glycemic Control
Brief Title: A Study to Test the Effectiveness and Safety of MK0893 in Combination With Other Drugs Used to Treat Type 2 Diabetes (0893-015)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0893-015; 2007_646
Record Dates: First submitted 2008-02-21; First posted 2008-03-07 (Estimated); Results first posted 2012-02-17 (Estimated); Last update posted 2017-01-02 (Estimated); Status verified 2016-12

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — N-((4-(1-(3-(3,5-dichlorophenyl)-5-(6-methoxynaphthalen-2-yl)-1H-pyrazol-1-yl)ethyl)phenyl)carbonyl)-beta-alanine; Sitagliptin Phosphate; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- MK-0893 + Sitagliptin (Experimental)
  Interventions: Drug: MK-0893; Drug: Sitagliptin; Drug: Placebo for Metformin
- MK-0893 + Metformin (Experimental)
  Interventions: Drug: MK-0893; Drug: Metformin; Drug: Placebo for Sitagliptin
- Sitagliptin + Metformin (Active Comparator)
  Interventions: Drug: Sitagliptin; Drug: Metformin; Drug: Placebo for MK-0893

INTERVENTIONS:
Drug: MK-0893 — Initial loading dose of 200 mg MK-0893 at randomization, followed by MK-0893 administered orally as 40 mg tablets daily throughout the double-blind treatment period (4 weeks).
  Arms: MK-0893 + Metformin; MK-0893 + Sitagliptin
Drug: Sitagliptin — Sitagliptin Phosphate administered orally as 100 mg tablets daily before the morning meal throughout the double-blind treatment period (4 weeks).
  Other Names: JANUVIA™; MK0431
  Arms: MK-0893 + Sitagliptin; Sitagliptin + Metformin
Drug: Metformin — Metformin taken orally (500 mg tablets) over an initial 2-week titration period starting at 500 mg administered twice daily before the morning and evening meals, increasing to 1500 mg daily, and ending with 1000 mg twice daily. Metformin then administered throughout the double-blind treatment period (4 weeks).
  Other Names: GLUCOPHAGE®
  Arms: MK-0893 + Metformin; Sitagliptin + Metformin
Drug: Placebo for MK-0893 — Matching placebo for MK-0893 was orally administered for the loading dose (200 mg) and for the following daily treatment (40 mg) over the 4 week double blind treatment period.
  Arms: Sitagliptin + Metformin
Drug: Placebo for Sitagliptin — Matching placebo for Sitagliptin (100 mg) administered orally as 100 mg tablets daily before the morning meal throughout the double-blind treatment period (4 weeks).
  Arms: MK-0893 + Metformin
Drug: Placebo for Metformin — Metformin-matched placebo taken orally (500 mg tablets) over an initial 2-week titration period starting at 500 mg administered twice daily before the morning and evening meals, increasing to 1500 mg daily, and ending with 1000 mg twice daily. Metformin-matched placebo then administered throughout the double-blind treatment period (4 weeks).
  Arms: MK-0893 + Sitagliptin

SUMMARY:
This study will test the effectiveness and safety of treatment with MK-0893 in combination with other drugs commonly used to treat type 2 diabetes for a duration up to 13 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have Type 2 Diabetes Mellitus, with suboptimal glucose control, while either not on AHA (antihyperglycemic agent) therapy or on monotherapy or on low-dose combination therapy

Exclusion Criteria:

* Participants have a history of Type 1 Diabetes Mellitus
* Participants taking insulin or thiazolidinediones (TZDs: peroxisome proliferator-activated receptor [PPAR]-gamma agonists)
* Participants who have a contraindication to metformin or sitagliptin

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2008-02; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants received matching placebos to MK-0893, Sitagliptin, and Metformin during a 2-week run-in period.
Groups:
- MK-0893 + Sitagliptin: Participants received an initial loading dose of 200 mg MK-0893 at randomization, followed by MK-0893 administered orally as 40 mg tablets daily throughout the double-blind treatment period. Sitagliptin was administered orally as 100 mg tablets daily before the morning meal throughout the double-blind treatment period.
- MK-0893 + Metformin: Participants received an initial loading dose of 200 mg MK-0893 at randomization, followed by MK-0893 orally (40 mg tablets) administered daily throughout the double-blind treatment period. Participants received Metformin orally (500 mg tablets) over an initial 2-week titration period starting at 500 mg administered twice daily before the morning and evening meals, increasing to 1500 mg daily, and ending with 1000 mg twice daily. Metformin was then administered throughout the double-blind treatment period.
- Sitagliptin + Metformin: Sitagliptin was administered orally as 100 mg tablets daily before the morning meal throughout the double-blind treatment period. Participants received Metformin orally (500 mg tablets) over an initial 2-week titration period starting at 500 mg administered twice daily before the morning and evening meals, increasing to 1500 mg daily, and ending with 1000 mg twice daily. Metformin was then administered throughout the double-blind treatment period.
Period: Overall Study
Arm/Group | MK-0893 + Sitagliptin | MK-0893 + Metformin | Sitagliptin + Metformin
Started | 48 | 49 | 49
Completed Post-Treatment Period | 44 | 47 | 47
Completed | 44 | 47 | 47
Not Completed | 4 | 2 | 2
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Lost to Follow-up | 2 | 2 | 0
Not completed — Physician Decision | 1 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MK-0893 + Sitagliptin | MK-0893 + Metformin | Sitagliptin + Metformin | Total
Number analyzed (Participants) | 48 | 49 | 49 | 146
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.6 (8.0) | 52.0 (9.7) | 53.8 (8.7) | 53.2 (8.8)
Gender [Count of Participants; unit: Participants]
  Female | 16 | 26 | 15 | 57
  Male | 32 | 23 | 34 | 89

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline (BL) to Week 4 in 24-hour Weighted Mean Glucose (WMG) Levels
Time Frame: BL, 4 weeks (end of double-blind treatment period)
Population: Full Analysis Set Population
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | MK-0893 + Sitagliptin | MK-0893 + Metformin | Sitagliptin + Metformin
Number analyzed (Participants) | 48 | 49 | 49
mg/dL | -85.7 (4.6) [4.6 to -117.4] | -117.4 (4.6) [-99.6 to 4.6] | -99.6 (4.6)
Statistical Analysis 1: Comparison: MK-0893 + Sitagliptin vs Sitagliptin + Metformin; Hypothesis: After 4 weeks of treatment, MK-0893+sitagliptin provide greater reduction in 24-hour WMG than sitagliptin+metformin. Using a standard deviation (SD) of 23.5 mg/dL, a sample size of 40 participants per group had 80% power to detect a true difference of 15 mg/dL in the mean change from BL in 24-hour WMG between any 2 treatment groups for a two-sided test at alpha=0.05, with a half-width of 10.3 mg/dL around the 95% confidence interval (CI) for the between group difference; Test type: Superiority or Other; p = 0.002, Longitudinal Data Analysis; Mean Difference (Final Values) = 13.9, 95% CI 2-sided [5.2 to 22.7]
Statistical Analysis 2: Comparison: MK-0893 + Metformin vs Sitagliptin + Metformin; Hypothesis: After 4 weeks of treatment, MK-0893+metformin provide greater reduction in 24-hour WMG than sitagliptin+metformin. Using a standard deviation (SD) of 23.5 mg/dL, a sample size of 40 participants per group had 80% power to detect a true difference of 15 mg/dL in the mean change from BL in 24-hour WMG between any 2 treatment groups for a two-sided test at alpha=0.05, with a half-width of 10.3 mg/dL around the 95% confidence interval for the between group difference; Test type: Superiority or Other; p < 0.001, Longitudinal Data Analysis; Mean Difference (Final Values) = -17.8, 95% CI 2-sided [-26.5 to -9.2]

2. Secondary Outcome: Change From BL to Week 4 in Fasting Plasma Glucose (FPG)
Time Frame: BL, 4 weeks (end of double-blind treatment period)
Population: Full Analysis Set Population
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | MK-0893 + Sitagliptin | MK-0893 + Metformin | Sitagliptin + Metformin
Number analyzed (Participants) | 48 | 49 | 49
mg/dL | -73.7 (4.4) | -101.9 (4.3) | -82.8 (4.3)
Statistical Analysis 1: Comparison: MK-0893 + Sitagliptin vs Sitagliptin + Metformin; Hypothesis: After 4 weeks of treatment, MK-0893+sitagliptin provide greater reduction in 24-hour FPG than sitagliptin+metformin. Using a standard deviation (SD) of 23.5 mg/dL, a sample size of 40 participants per group had 80% power to detect a true difference of 15 mg/dL in the mean change from BL in 24-hour FPG between any 2 treatment groups for a two-sided test at alpha=0.05, with a half-width of 10.3 mg/dL around the 95% confidence interval for the between group difference; Test type: Superiority or Other; p = 0.050, Longitudinal Data Analysis; Mean Difference (Final Values) = 9.1, 95% CI 2-sided [0.0 to 18.2]
Statistical Analysis 2: Comparison: MK-0893 + Metformin vs Sitagliptin + Metformin; Hypothesis: After 4 weeks of treatment, MK-0893+metformin provide greater reduction in 24-hour FPG than sitagliptin+metformin. Using a standard deviation (SD) of 23.5 mg/dL, a sample size of 40 participants per group had 80% power to detect a true difference of 15 mg/dL in the mean change from BL in 24-hour FPG between any 2 treatment groups for a two-sided test at alpha=0.05, with a half-width of 10.3 mg/dL around the 95% confidence interval for the between group difference; Test type: Superiority or Other; p < 0.001, Longitudinal Data Analysis; Mean Difference (Final Values) = -19.1, 95% CI 2-sided [-28.0 to -10.1]

3. Secondary Outcome: Change From BL to Week 4 in 2-hr Glucose Area Under The Curve (AUC)
Time Frame: BL, 4 weeks (end of double-blind treatment period)
Population: Full Analysis Set Population
Measure: Least Squares Mean (Standard Error); unit: mg.h/dL
Arm/Group | MK-0893 + Sitagliptin | MK-0893 + Metformin | Sitagliptin + Metformin
Number analyzed (Participants) | 48 | 49 | 49
mg.h/dL | -187.7 (11.4) | -254.9 (11.1) | -210.3 (11.4)
Statistical Analysis 1: Comparison: MK-0893 + Sitagliptin vs Sitagliptin + Metformin; Hypothesis: After 4 weeks of treatment, MK-0893+sitagliptin provide greater reduction in 2-hr Glucose AUC than sitagliptin+metformin. Using a SD of 23.5 mg/dL, a sample size of 40 participants per group had 80% power to detect a true difference of 15 mg/dL in the mean change from BL in 2-Hour Glucose Total AUC between any 2 treatment groups for a two-sided test at alpha=0.05, with a half-width of 10.3 mg/dL around the 95% confidence interval for the between group difference; Test type: Superiority or Other; p = 0.056, Longitudinal Data Analysis; Mean Difference (Final Values) = 22.6, 95% CI 2-sided [-0.6 to 45.8]
Statistical Analysis 2: Comparison: MK-0893 + Metformin vs Sitagliptin + Metformin; Hypothesis: After 4 weeks of treatment, MK-0893+metformin provide greater reduction in 2-hr Glucose AUC than sitagliptin+metformin. Using a SD of 23.5 mg/dL, a sample size of 40 participants per group had 80% power to detect a true difference of 15 mg/dL in the mean change from BL in 2-Hour Glucose Total AUC between any 2 treatment groups for a two-sided test at alpha=0.05, with a half-width of 10.3 mg/dL around the 95% confidence interval for the between group difference; Test type: Superiority or Other; p < 0.001, Longitudinal Data Analysis; Mean Difference (Final Values) = -44.6, 95% CI 2-sided [-67.3 to -21.8]

4. Secondary Outcome: Change From BL to Week 4 in the 2-Hour Total GLP-1 Total AUC
Description: Glucagon-Like Peptide-1 (GLP-1) is an incretin hormone that acts as a potent insulin secretegogue in response to nutrient ingestion and stimulates glucose disposition. The total AUC of Total GLP-1 levels was calculated from blood sample data measured after the morning meal.
Time Frame: BL, 4 weeks (end of double-blind treatment period)
Population: Full Analysis Set Population
Measure: Least Squares Mean (Standard Error); unit: pmol*h/L
Arm/Group | MK-0893 + Sitagliptin | MK-0893 + Metformin | Sitagliptin + Metformin
Number analyzed (Participants) | 48 | 49 | 49
pmol*h/L | 7.4 (1.0) | 16.4 (1.0) | 3.2 (1.0)
Statistical Analysis 1: Comparison: MK-0893 + Sitagliptin vs Sitagliptin + Metformin; Hypothesis: After 4 weeks of treatment, MK-0893+sitagliptin provide greater reduction in 2-Hour Total GLP-1 Total AUC than sitagliptin+metformin. Using a SD of 23.5 mg/dL, a sample size of 40 participants/group had 80% power to detect a true difference of 15 mg/dL in the mean change from BL in 2-Hour Total GLP-1 Total AUC between any 2 treatment groups for a 2-sided test at alpha=0.05, with a half-width of 10.3 mg/dL around the 95% CI for the between group difference; Test type: Superiority or Other; p = 0.001, Longitudinal Data Analysis; Mean Difference (Final Values) = 4.2, 95% CI 2-sided [1.7 to 6.7]
Statistical Analysis 2: Comparison: MK-0893 + Metformin vs Sitagliptin + Metformin; Hypothesis: After 4 weeks of treatment, MK-0893+metformin provide greater reduction in 2-Hour Total GLP-1 Total AUC than sitagliptin+metformin. Using a SD of 23.5 mg/dL, a sample size of 40 participants/group had 80% power to detect a true difference of 15 mg/dL in the mean change from BL in 2-Hour Total GLP-1 Total AUC between any 2 treatment groups for a 2-sided test at alpha=0.05, with a half-width of 10.3 mg/dL around the 95% CI for the between group difference; Test type: Superiority or Other; p < 0.001, Longitudinal Data Analysis; Mean Difference (Final Values) = 13.2, 95% CI 2-sided [10.7 to 15.7]

5. Secondary Outcome: Change From BL to Week 4 in the 2-Hour Active GLP-1 Total AUC
Description: GLP-1 is cleaved from proglucagon to form the active peptide GLP-1. The active form promotes suppression of glucagon secretion. The total AUC of Active GLP-1 levels was calculated from blood sample data measured after the morning meal.
Time Frame: BL, 4 weeks (end of double-blind treatment period)
Population: Full Analysis Set Population
Measure: Least Squares Mean (Standard Error); unit: pmole*h/L
Arm/Group | MK-0893 + Sitagliptin | MK-0893 + Metformin | Sitagliptin + Metformin
Number analyzed (Participants) | 48 | 49 | 49
pmole*h/L | 11.0 (1.1) | 6.3 (1.1) | 17.6 (1.1)
Statistical Analysis 1: Comparison: MK-0893 + Sitagliptin vs Sitagliptin + Metformin; Hypothesis: After 4 weeks of treatment, MK-0893+sitagliptin provide greater reduction in 2-Hour Active GLP-1 Total AUC than sitagliptin+metformin. Using a SD of 23.5 mg/dL, a sample size of 40 participants/group had 80% power to detect a true difference of 15 mg/dL in the mean change from BL in 2-Hour Active GLP-1 Total AUC between any 2 treatment groups for a 2-sided test at alpha=0.05, with a half-width of 10.3 mg/dL around the 95% CI for the between group difference; Test type: Superiority or Other; p < 0.001, Longitudinal Data Analysis; Mean Difference (Final Values) = -6.7, 95% CI 2-sided [-9.5 to -3.8]
Statistical Analysis 2: Comparison: MK-0893 + Metformin vs Sitagliptin + Metformin; Hypothesis: After 4 weeks of treatment, MK-0893+metformin provide greater reduction in 2-Hour Active GLP-1 Total AUC than sitagliptin+metformin. Using a SD of 23.5 mg/dL, a sample size of 40 participants/group had 80% power to detect a true difference of 15 mg/dL in the mean change from BL in 2-Hour Active GLP-1 Total AUC between any 2 treatment groups for a 2-sided test at alpha=0.05, with a half-width of 10.3 mg/dL around the 95% CI for the between group difference; Test type: Superiority or Other; p < 0.001, Longitudinal Data Analysis; Mean Difference (Final Values) = -11.3, 95% CI 2-sided [-14.1 to -8.5]

ADVERSE EVENTS:
Arm/Group | MK-0893 + Sitagliptin | MK-0893 + Metformin | Sitagliptin + Metformin
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/49 | 0/49
Other Adverse Events (participants affected / at risk) | 7/48 | 10/49 | 8/49
OTHER ADVERSE EVENTS (reported when occurring in more than 5.0% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-0893 + Sitagliptin (N=48) | MK-0893 + Metformin (N=49) | Sitagliptin + Metformin (N=49)
diarrhoea (Gastrointestinal disorders) | 1 (1) | 6 (7) | 6 (9)
nausea (Gastrointestinal disorders) | 2 (2) | 4 (5) | 2 (2)
upper respiratory tract infection (Infections and infestations) | 4 (4) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission. SPONSOR review can be expedited to meet publication guidelines.